CLINICAL TRIAL: NCT02401464
Title: A Randomized, Open-label, 2×2 Crossover, Phase I Study to Evaluate the Bioequivalence of Single Oral Dose of TAK-536 Pediatric Formulations and TAK-536 Commercial Tablet in Healthy Adult Male Subjects
Brief Title: A Bioequivalence Study of TAK-536 Pediatric Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-536/CPH-101; U1111-1168-3113 (Registry Identifier: WHO); JapicCTI-152853 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-05

CONDITIONS: Japanese Healthy Adult Males
MeSH Terms: interventions — azilsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dry syrup formulation (Group a) (Experimental): One pack of the dry syrup formulation of TAK-536, containing 10 milligram (mg) of TAK-536, will be orally administered with water (200 milliliter [mL]) at breakfast to fasting participants who have fasted for 10 hours or longer since the night prior to the administration of study medication in Period 1 and, after a washout period of 6 days or more, one 10 mg tablet of TAK-536 will be orally administered with water (200 mL) at breakfast to fasting participants who have fasted for 10 hours or longer since the night prior to the administration of study medication in Period 2.
  Interventions: Drug: TAK-536 Tablet; Drug: TAK-536 Dry Syrup Formulation
- Dry syrup formulation (Group b) (Experimental): One 10 mg tablet of TAK-536 will be orally administered with water (200 mL) at breakfast to fasting participants who have fasted for 10 hours or longer since the night prior to the administration of study medication in Period 1 and, after a washout period of 6 days or more, one pack of the dry syrup formulation of TAK-536, containing 10 mg of TAK-536, will be orally administered with water (200 mL) at breakfast to fasting participants who have fasted for 10 hours or longer since the night prior to the administration of study medication in Period 2.
  Interventions: Drug: TAK-536 Tablet; Drug: TAK-536 Dry Syrup Formulation
- Granule formulation (Group a) (Experimental): One pack of the granule formulation of TAK-536, containing 10 mg of TAK-536,will be orally administered with water (200 mL) at breakfast to fasting participants who have fasted for 10 hours or longer since the night prior to the administration of study medication in Period 1 and, after a washout period of 6 days or more, one 10 mg tablet of TAK-536 will be orally administered with water (200 mL) at breakfast to fasting participants who have fasted for 10 hours or longer since the night prior to the administration of study medication in Period 2.
  Interventions: Drug: TAK-536 Tablet; Drug: TAK-536 Ganule Formulation
- Granule formulation (Group b) (Experimental): One 10 mg tablet of TAK-536 will be orally administered with water (200 mL) at breakfast to fasting participants who have fasted for 10 hours or longer since the night prior to the administration of study medication in Period 1 and, after a washout period of 6 days or more, one pack of the granule formulation of TAK-536, containing 10 mg of TAK-536, will be orally administered with water (200 mL) at breakfast to fasting participants who have fasted for 10 hours or longer since the night prior to the administration of study medication in Period 2.
  Interventions: Drug: TAK-536 Tablet; Drug: TAK-536 Ganule Formulation

INTERVENTIONS:
Drug: TAK-536 Tablet — TAK-536 10 mg tablet
Drug: TAK-536 Dry Syrup Formulation — TAK-536 dry syrup formulation
  Arms: Dry syrup formulation (Group a); Dry syrup formulation (Group b)
Drug: TAK-536 Ganule Formulation — TAK-536 granule formulation
  Arms: Granule formulation (Group a); Granule formulation (Group b)

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of a single oral dose of 2 different drug forms of TAK-536 pediatric formulation and a single oral dose of TAK-536 commercial tablet in healthy Japanese adult male participants.

DETAILED DESCRIPTION:
This study was designed to evaluate the bioequivalence of a single oral dose of 2 different drug forms of TAK-536 pediatric formulation (dry syrup, granules) and a single oral dose of TAK-536 commercial tablet by using open-label, 2 × 2 crossover design.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or the sub-investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form (ICF) and any required privacy authorization prior to the initiation of any study procedures.
3. The participant is a healthy Japanese adult male volunteer.
4. The participant is between 20 and 35 years of age at the time of informed consent.
5. The participant has a body weight of at least 50.0 kilogram (kg) and has a body mass index (BMI) between 18.5 and 25.0 kilogram per meter square (kg/m^2) at the time of screening.

Exclusion Criteria:

1. The participant has shown symptoms of dizziness on standing up, facial pallor, cold sweat, etc, and suspected hypotension at medical examination/physical findings at screening and the day before administration of the study drug for Period 1, and before administration of the study drug for Period 1.
2. The participant has received any investigational compound within 16 weeks (112 days) prior to the start of study medication for Period 1
3. The participant has received TAK-536 or TAK-491 in a previous clinical study or as a therapeutic agent.
4. The participant has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic or endocrine disease or other abnormality which may impact the ability of the participant to participate or potentially confound the study results.
5. The participant has a known hypersensitivity to TAK-536 or angiotensin II receptor blockers.
6. The participant has positive results in the urine drug screening test at screening.
7. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to the screening or is unwilling to agree to abstain from alcohol and drugs throughout the study period.
8. The participant has taken any excluded medication, supplements, or food products during the time periods.
9. The participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention (ie, cholecystectomy).
10. The participant has a history of cancer.
11. The participant has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen, or serological reactions for syphilis at screening.
12. The participant has poor peripheral venous access.
13. The participant has undergone whole blood collection of at least 200 mL within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to the start of study medication administration for Period 1.
14. The participant has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to the start of study medication administration for Period 1.
15. The participant has undergone blood component collection within 2 weeks (14 days) prior to the start of study medication administration for Period 1.
16. The participant has an abnormal (clinically significant) electro-cardiogram at screening or prior to the start of study medication for Period 1.
17. The participant has abnormal laboratory values at screening or prior to the start of study medication for Period 1 that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine transaminase (ALT) or aspartate transaminase (AST) greater than (>)1.5 times the upper limits of normal.
18. The participant who, in the opinion of the investigator or the sub-investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Kagoshima, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 25 March 2015 to 26 May 2015.
Pre-assignment Details: Healthy participants were enrolled in 1 of 2 treatment sequences: Sequence a (dry syrup): TAK-536 dry syrup followed by TAK-536 tablet; Sequence b (dry syrup): TAK-536 tablet followed by TAK-536 dry syrup; Sequence a (granules): TAK-536 granules followed by TAK-536 tablet; Sequence b (granules): TAK-536 tablet followed by TAK-536 granules.
Groups:
- Dry Syrup Cohort: TAK-536 Dry Syrup + TAK-536 Tablet: Participants in Sequence a of dry syrup formulation received TAK-536 10 milligram (mg), dry syrup (pediatric formulation), orally, once on Day 1 of Intervention Period 1 (6 days), followed by washout period of at least 6 days, further followed by TAK-536 10 mg, tablet (commercial formulation), orally, once on Day 1 of Intervention Period 2 (6 days).
- Dry Syrup Cohort: TAK-536 Tablet + TAK-536 Dry Syrup: Participants in Sequence b of dry syrup formulation received TAK-536 10 mg, tablet (commercial formulation), orally, once on Day 1 of Intervention Period 1 (6 days), followed by washout period of at least 6 days, further followed by TAK-536 10 mg, dry syrup (pediatric formulation), orally, once on Day 1 of Intervention Period 2 (6 days).
- Granule Cohort: TAK-536 Granules + TAK-536 Tablet: Participants in Sequence a of granules formulation received TAK-536 10 mg, granules (pediatric formulation), orally, once on Day 1 of Intervention Period 1 (6 days), followed by washout period of at least 6 days, further followed by TAK-536 10 mg, tablet (commercial formulation), orally, once on Day 1 of Intervention Period 2 (6 days).
- Granule Cohort: TAK-536 Tablet + TAK-536 Granules: Participants in Sequence b of granules formulation received TAK-536 10 mg, tablet (commercial formulation), orally, once on Day 1 of Intervention Period 1 (6 days) followed by washout period of at least 6 days, further followed by TAK-536 10 mg, granules (pediatric formulation), orally, once on Day 1 of Intervention Period 2 (6 days).
Period: Intervention Period 1 (6 Days)
Arm/Group | Dry Syrup Cohort: TAK-536 Dry Syrup + TAK-536 Tablet | Dry Syrup Cohort: TAK-536 Tablet + TAK-536 Dry Syrup | Granule Cohort: TAK-536 Granules + TAK-536 Tablet | Granule Cohort: TAK-536 Tablet + TAK-536 Granules
Started | 13 | 13 | 13 | 13
Completed | 13 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (At Least 6 Days)
Arm/Group | Dry Syrup Cohort: TAK-536 Dry Syrup + TAK-536 Tablet | Dry Syrup Cohort: TAK-536 Tablet + TAK-536 Dry Syrup | Granule Cohort: TAK-536 Granules + TAK-536 Tablet | Granule Cohort: TAK-536 Tablet + TAK-536 Granules
Started | 13 | 13 | 13 | 13
Completed | 13 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Intervention Period 2 (6 Days)
Arm/Group | Dry Syrup Cohort: TAK-536 Dry Syrup + TAK-536 Tablet | Dry Syrup Cohort: TAK-536 Tablet + TAK-536 Dry Syrup | Granule Cohort: TAK-536 Granules + TAK-536 Tablet | Granule Cohort: TAK-536 Tablet + TAK-536 Granules
Started | 13 | 13 | 13 | 13
Completed | 13 | 13 | 13 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The pharmacokinetic analysis set included all participants who received the study drug, completed the minimum protocol-specified procedures without any major protocol deviations, and were evaluable for pharmacokinetics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dry Syrup Cohort: TAK-536 Dry Syrup + TAK-536 Tablet | Dry Syrup Cohort: TAK-536 Tablet + TAK-536 Dry Syrup | Granule Cohort: TAK-536 Granules + TAK-536 Tablet | Granule Cohort: TAK-536 Tablet + TAK-536 Granules | Total
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (2.21) | 25.9 (4.11) | 26.6 (4.07) | 27.4 (5.71) | 26.308 (4.16)
Sex/Gender, Customized [Number; unit: participants]
  Male | 13 | 13 | 13 | 13 | 52
Smoking classification [Number; unit: participants]
  Never smoked | 7 | 9 | 7 | 8 | 31
  Current smoker | 0 | 0 | 1 | 1 | 2
  Ex-smoker | 6 | 4 | 5 | 4 | 19
Alcohol classification [Number; unit: participants]
  Drank a few days per week | 1 | 2 | 2 | 0 | 5
  Drank a few days per month | 1 | 3 | 3 | 3 | 10
  Never drank | 11 | 8 | 8 | 10 | 37
Caffeine Classification [Number; unit: participants]
  Had caffeine consumption | 2 | 3 | 6 | 5 | 16
  Had no caffeine consumption | 11 | 10 | 7 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-48): Area Under the Plasma Concentration-Time Curve From Time 0 to 48 Hours Postdose for TAK-536 in Dry Syrup Cohort
Time Frame: Day 1: pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation: Participants received TAK-536 10 mg, dry syrup (pediatric formulation), orally, once on Day 1 of either Intervention Period 1 or 2 (6 days).
- Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation: Participants received TAK-536 10 mg, tablet (commercial formulation), orally, once on Day 1 of Intervention Period 1 or 2 (6 days).
Arm/Group | Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation | Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation
Number analyzed (Participants) | 26 | 26
nanogram*hour per milliliter (ng*hr/mL) | 7065.6 (1317.91) | 7341.2 (1493.71)
Statistical Analysis 1: Comparison: Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation vs Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation; Based on the analysis of variance (ANOVA) in which the natural logarithms of AUC(0-48) of TAK-536 were used as dependent variables, and formulation, sequence (administration order) and administration period were used as fixed effects, bioequivalence was assessed providing two-sided 90% confidence intervals (CIs) for the differences between the formulations and between the periods; Test type: Non-Inferiority or Equivalence — Formulations were considered bioequivalent if: 1) 90% Cls of the differences in the means of the natural log-transformed AUC(0-48) and Cmax between commercial and pediatric formulations was within ln(0.80)- ln(1.25);2) Differences in the means of the natural log-transformed AUC(0-48) and Cmax between commercial and pediatric formulations was within ln(0.9)-ln(1.11),and results of the dissolution test met the conditions specified in the Guideline for Bioequivalence Studies of Generic Products; Least Squares (LS) mean difference (ln) = 0.963, 90% CI 2-sided [0.927 to 1.001]

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-536 in Dry Syrup Cohort
Time Frame: Day 1: pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation | Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation
Number analyzed (Participants) | 26 | 26
nanogram per milliliter (ng/mL) | 886.1 (133.76) | 976.7 (140.97)
Statistical Analysis 1: Comparison: Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation vs Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation; Based on the ANOVA in which the natural logarithms of Cmax of TAK-536 were used as dependent variables, and formulation, sequence (administration order) and administration period were used as fixed effects, bioequivalence was assessed providing two-sided 90% CIs for the differences between the formulations and between the periods; Test type: Non-Inferiority or Equivalence — Formulations were considered bioequivalent if: 1)90% Cls of the differences in the means of the natural log-transformed AUC(0-48) and Cmax between commercial and pediatric formulations was within ln(0.80)- ln(1.25);2) Differences in the means of the natural log-transformed AUC(0-48) and Cmax between commercial and pediatric formulations was within ln(0.9)-ln(1.11),and results of the dissolution test met the conditions specified in the Guideline for Bioequivalence Studies of Generic Products; LS mean difference (ln) = 0.906, 90% CI 2-sided [0.880 to 0.933]

3. Primary Outcome: AUC(0-48): Area Under the Plasma Concentration-Time Curve From Time 0 to 48 Hours Postdose for TAK-536 in Granule Cohort
Time Frame: Day 1: pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Granule Cohort: TAK-536 10 mg Pediatric Formulation: Participants received TAK-536 10 mg, granule (pediatric formulation), orally, once on Day 1 of Intervention Period 1 or 2 (6 days).
- Granule Cohort: TAK-536 10 mg Commercial Formulation: Participants received TAK-536 10 mg, tablet (commercial formulation), orally, once on Day 1 of Intervention Period 1 or 2 (6 days).
Arm/Group | Granule Cohort: TAK-536 10 mg Pediatric Formulation | Granule Cohort: TAK-536 10 mg Commercial Formulation
Number analyzed (Participants) | 26 | 26
ng*hr/mL | 7749.8 (1188.80) | 7893.2 (1336.61)
Statistical Analysis 1: Comparison: Granule Cohort: TAK-536 10 mg Pediatric Formulation vs Granule Cohort: TAK-536 10 mg Commercial Formulation; Based on the ANOVA in which the natural logarithms of AUC(0-48) of TAK-536 were used as dependent variables, and formulation, sequence (administration order) and administration period were used as fixed effects, bioequivalence was assessed providing two-sided 90% CIs for the differences between the formulations and between the periods; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; LS mean difference (ln) = 0.985, 90% CI 2-sided [0.958 to 1.011]

4. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-536 in Granule Cohort
Time Frame: Day 1: pre-dose and at multiple timepoints (up to 48 hours) post-dose
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Granule Cohort: TAK-536 10 mg Pediatric Formulation | Granule Cohort: TAK-536 10 mg Commercial Formulation
Number analyzed (Participants) | 26 | 26
ng/mL | 943.2 (106.76) | 973.7 (178.75)
Statistical Analysis 1: Comparison: Granule Cohort: TAK-536 10 mg Pediatric Formulation vs Granule Cohort: TAK-536 10 mg Commercial Formulation; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; LS mean difference (ln) = 0.979, 90% CI 2-sided [0.938 to 1.022]

5. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to Day 6 of Intervention Period 2
Population: The safety analysis set included all participants who received the study drug at least once.
Measure: Number; unit: participants
Arm/Group | Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation | Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation | Granule Cohort: TAK-536 10 mg Pediatric Formulation | Granule Cohort: TAK-536 10 mg Commercial Formulation
Number analyzed (Participants) | 26 | 26 | 26 | 26
participants | 5 | 5 | 0 | 3

6. Secondary Outcome: Number of Participants With TEAEs Related to Vital Signs
Time Frame: Baseline up to Day 6 of Intervention Period 2
Population: The safety analysis set included all participants who received the study drug at least once.
Measure: Number; unit: participants
Arm/Group | Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation | Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation | Granule Cohort: TAK-536 10 mg Pediatric Formulation | Granule Cohort: TAK-536 10 mg Commercial Formulation
Number analyzed (Participants) | 26 | 26 | 26 | 26
participants | 0 | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With TEAEs Related to Body Weight
Time Frame: Baseline up to Day 6 of Intervention Period 2
Population: The safety analysis set included all participants who received the study drug at least once.
Measure: Number; unit: participants
Arm/Group | Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation | Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation | Granule Cohort: TAK-536 10 mg Pediatric Formulation | Granule Cohort: TAK-536 10 mg Commercial Formulation
Number analyzed (Participants) | 26 | 26 | 26 | 26
participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Who Had Clinically Meaningful Changes From Baseline in 12-lead Electrocardiograms (ECG)
Time Frame: Baseline up to Day 6 of Intervention Period 2
Population: The safety analysis set included all participants who received the study drug at least once.
Measure: Number; unit: participants
Arm/Group | Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation | Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation | Granule Cohort: TAK-536 10 mg Pediatric Formulation | Granule Cohort: TAK-536 10 mg Commercial Formulation
Number analyzed (Participants) | 26 | 26 | 26 | 26
participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With TEAEs Categorized Into Investigations System Organ Class (SOC) Related to Laboratory Values
Time Frame: Baseline up to Day 6 of Intervention Period 2
Population: The safety analysis set included all participants who received the study drug at least once.
Measure: Number; unit: participants
Arm/Group | Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation | Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation | Granule Cohort: TAK-536 10 mg Pediatric Formulation | Granule Cohort: TAK-536 10 mg Commercial Formulation
Number analyzed (Participants) | 26 | 26 | 26 | 26
participants | 4 | 5 | 0 | 2

ADVERSE EVENTS:
Time Frame: Collection of AEs commenced from the time that the participant was first administered study drug in Period 1 (Baseline) and continued until the follow-up examination in Period 2 (Day 6 of Intervention Period 2).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation | Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation | Granule Cohort: TAK-536 10 mg Pediatric Formulation | Granule Cohort: TAK-536 10 mg Commercial Formulation
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 5/26 | 5/26 | 0/26 | 3/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dry Syrup Cohort: TAK-536 10 mg Pediatric Formulation (N=26) | Dry Syrup Cohort: TAK-536 10 mg Commercial Formulation (N=26) | Granule Cohort: TAK-536 10 mg Pediatric Formulation (N=26) | Granule Cohort: TAK-536 10 mg Commercial Formulation (N=26)
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Protein urine present (Investigations) | 2 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.